CLINICAL TRIAL: NCT01022398
Title: Vitamin D Replacement: The Effect on Statin-Related Myalgias
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment slow, funding ended.
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-15532
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2012-09

CONDITIONS: HMG-CoA Reductase Inhibitors-related Myalgias
Keywords: Vitamin D3; HMG-CoA reductase inhibitors (statin)-related myalgias
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): Subjects will receive Vitamin D supplementation 10,000 international units of cholecalciferol (vitamin D3) by mouth weekly
  Interventions: Drug: cholecalciferol/placebo
- Placebo (Placebo Comparator): Subjects will receive placebo (an exact replica of the vitamin D capsule that does not contain any medically active substance) by mouth weekly
  Interventions: Drug: cholecalciferol/placebo

INTERVENTIONS:
Drug: cholecalciferol/placebo — 10,000 IU by mouth weekly for 6 months
  Other Names: Vitamin D3/placebo

SUMMARY:
The purpose of this project is to determine if Vitamin D supplementation [10,000 international units of cholecalciferol (vitamin D3) by mouth weekly] will decrease the rate of discontinuation of statin therapy due to muscle ache/pain and decrease the occurrence of muscle ache/pain due to statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who recently prescribed statins (in the last seven days) or who have had a recent increase in statin dose (in the last seven days)
* Patients aged 19-89 years old
* Men and women (not of childbearing potential)
* Patients receiving statins with concomitant ezetimibe

Exclusion Criteria:

* history of alcoholism or malnutrition
* receiving concomitant niacin, fibric acid derivatives, bile acid sequestrants, or other drugs that affect cholesterol levels

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Schima, MD, Principal Investigator — Creighton University
Locations (1):
- The Cardiac Center at Creighton University, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Study terminated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (1.4) | 56.5 (16.2) | 52.75 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Determine if the Replacement of Vitamin D 10,000 IU Weekly Will Decrease the Discontinuation Rate of Statin Therapy and Decrease the Incidence of Statin-related Myalgia in Patients Requiring Statin Therapy
Time Frame: 6 months
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Adverse Events Not Collected: Adverse Events Not Collected
Arm/Group | Adverse Events Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes